CLINICAL TRIAL: NCT07290907
Title: EFFECTIVENESS OF HOME-BASED CARDIAC REHABILITATION TO IMPROVE QUALITY OF LIFE AND HEALTH BEHAVIOR OF PATIENTS WITH CARDIOVASCULAR DISEASES IN LOW-RESOURCE SETTINGS IN PAKISTAN
Brief Title: Effectiveness of Home-Based Cardiac Rehabilitation
Acronym: NCD CVD HBCR
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Pakistan Institute of Medical Sciences (Other Government)
Responsible Party: Principal Investigator, Liaquat Ali, Assistant Clinical Instructor, Pakistan Institute of Medical Sciences
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: F-5-2/2024 ERRC
Record Dates: First submitted 2025-12-03; First posted 2025-12-18 (Actual); Last update posted 2025-12-18 (Actual); Status verified 2025-12

CONDITIONS: Cardiac Rehabilitation

STUDY DESIGN:
Intervention Model Description: The control group will receive only standard communication from the cardiologist and routine follow-up care. The control group will receive standard discharge advice and routine outpatient follow-up care as per hospital protocol, with no structured rehabilitation support. Home-based cardiac rehabilitation for the intervention group will be supervised by a multidisciplinary team such as a researcher, trained nursing staff, and cardiologist. A structured cardiac rehabilitation program will be conducted at the patient's home. This structured program will include dietary counseling, physical activity suggestions and recommendations, adherence to medications prescribed by the cardiologist, psychotherapy, and lastly telephone calls or visits at home. The time duration of the data collection will start from the baseline to the intervention, comprising 12 weeks.
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- The Intervention group (Cardiac Rehabilitation Program) (Experimental): The Intervention group Home-based cardiac rehabilitation for the intervention group. A structured cardiac rehabilitation program will be conducted at the patient's home. This structured program will include dietary counseling, physical activity suggestions and recommendations, adherence to medications prescribed by the cardiologist, psychotherapy, and lastly telephone calls or visits at home.
  Interventions: Behavioral: Home-based therapy
- Control group (No Intervention): The control group will receive only standard communication from the cardiologist and routine follow-up care. The control group will receive standard discharge advice and routine outpatient follow-up care as per hospital protocol, with no structured rehabilitation support.

INTERVENTIONS:
Behavioral: Home-based therapy — A structured cardiac rehabilitation program will be conducted at the patient's home. This structured program will include dietary counseling, physical activity suggestions and recommendations, adherence to medications prescribed by the cardiologist, psychotherapy, and lastly telephone calls or visits at home.
  Arms: The Intervention group (Cardiac Rehabilitation Program)

SUMMARY:
Statement of the Problem WHO stated that the average life expectancy has been recorded as 40 years among these in South Asian countries and 98 million people relate to Pakistan. Wang pointed out that the significant difference has been seen regarding provision of the health care facilities being provided in the rural and urban settings, called as health poverty in rural area as compared to urban areas. Therefore, accessibility of essential healthcare facilities such as experienced staff, vaccination and necessarily supply of medicines in rural population would be supporting reducing health poverty and will maintain equal and equitable opportunities. Andersen and Newman argued that there are main factors such as distance, time and travel costs that affect health accessibility for the poor people living in rural settings which are deprived of emergency care and common in developing economies.

Cardiac Rehabilitation is a efficient, safe and affordable intervention that lowers overall health service financial burden. Additionally, CR are planned to optimize and restore physical, psychological, and social functioning by combining medical consultation, individualized exercise sessions, education, cardiac risk factor modification, and health counseling. CR is highly and mostly suggested as the key multicomponent and multi-dimensional intervention for the prevention of death by cardiac attacks, the lowering chances of hospital readmissions, and the enhancement of quality of life (QoL) of the people. Therefore, CR is one of the effective techniques to decrease the increasing number of cases and provide an efficient cardiac health intervention program with appropriate planning and organization.

Despite the evidence of cost-effective rehabilitation program to optimize cardiac functioning at the hospital-based settings but the participation in cardiac rehabilitation, traditionally delivered in hospital outpatient departments or community, Despite the evidence of cost-effective rehabilitation program to optimize cardiac functioning at the hospital-based settings but the participation in cardiac rehabilitation, traditionally delivered in hospital outpatient departments or community centers, has remained low, with average participation rates < 20% recorded in the United States and similarly in the Europe. Low participation has predominantly recorded mostly in few groups like women, elder population, ethnic minorities, and those living in rural settings or who are socioeconomically and financially resource constrained. Subsequently, these patients were contacted through calls for alternative options to center-based cardiac rehabilitation. Recommended interventions included cardiac rehabilitation at home transited by healthcare professionals with the support of telehealth technologies to maximize participation. Thus, the home-based cardiac rehabilitation program was recommended by the American Heart Association and the American College of Cardiology in 2019 through a scientific statement. Guidelines from NICE on chronic heart failure in the UK in 2018 said that "delivery of home-based rehabilitation may enhance the accessibility and participation. For changing behavior and improving quality of life, HBCR is an essential component of secondary prevention and an important alternative technique, for those patients who suffered a cardiac incident or experienced any other cardiac event. Hence, HBCR is one of the effective t strategies to reduce the higher number of cases. HBCR contains techniques for secondary prevention that facilitate cardiac patients to rebuild their functional cardiac capacity and decrease the magnitude of hospital visits and workload in emergency management in coronary critical areas.

Most of the studies were done on cardiovascular disease and on the conventional approach of hospital-based cardiac rehabilitation, but rare literature in the context of Pakistan, especially Islamabad, was found on home-based cardiac rehabilitation to improve the quality of life and behavior of the patients. Thus, the study aims to evaluate the effectiveness of home-based cardiac rehabilitation to improve the quality of life and health behavior of patients with cardiovascular disease in low resource settings in Islamabad.

DETAILED DESCRIPTION:
Objectives of Study H01: There is a significant difference in the quality of life and health behavior of patients with cardiovascular diseases who will receive usual care with and without HBCR.

H02: There is a significant difference in the frequency of emergency hospital visits of patients with cardiovascular diseases who will receive usual care with and without HBCR Significance of Study Benefits for the Development of Knowledge This research has the potential to provide significant contributions to the development of the knowledge in the field of health sector specially nursing and cardiology and public health. This study may encourage the development of the Home based cardiac rehabilitation and may encourage to provide accessible and affordable health care services. Home-based cardiac rehabilitation (HBCR) is a research-based intervention to improve quality of life and health behavior, preventing cardiovascular diseases. It will be significant, as its findings will bring results to improve home-based nursing care for the improvement of life and behavior of cardiac patients. Besides, this research enhances the comprehensive strategy to understand the differences and similarities in applying HBCR model in various cultures and regions.

Benefits to the Community This study provides direct benefits to the community especially to rural health of how resource settings which need awareness, cost effective, accessible and affordable health care services. Families and patients will be able to manage their cardiac health by controlling risk factors and changing life styles that affect cardiac health.

Benefits for Policymakers This research will be able to provide opportunity to policy makers at local and regional level to devise strategies and policies based on scientific evidence to provide cardiac health care services to the low resource settings. The results of this study will also be shared with key stakeholders associated with nursing and health policy-making subjects, such as the Pakistan Nursing & Midwifery Council and health ministry at the national and provincial levels. This will help in identifying the needs that could meet the standards and protocols of home-based cardiac rehabilitation and changes in curriculum of nursing education focusing cardiac health.

Benefits to the Country Home based Cardiac rehabilitation will improve quality of life and reduce healthcare expenditure burden of the country. The exercise component of the intervention of HBCR will provide significant physiological positive outcomes, including increased maximal oxygen uptake (VO2 max), normal endothelial functioning, and improved myocardial capability to function. Besides, cardiac rehabilitation will help in reductions in smoking, lowering body weight, improving serum lipids, and blood pressure. A Cochrane review found that cardiac rehabilitation reduced hospital admissions and impacted to a long-term reduction in all-cause mortality in patients with heart failure and preserved ejection fraction, though no short-term (<12 months) mortality benefit was observed. Besides, reduced burden of admissions and expenditure on the hospital.

Scope of Study This research study is conducted to evaluate the effectiveness of home-based cardiac rehabilitation to improve the quality of life and health behavior of patients with cardiovascular disease in low-resource settings in Islamabad, Pakistan. Patients diagnosed with cardiovascular disease will be included as the target population in this study. The scope of this study will be to analyze the effectiveness of home-based cardiac rehabilitation to improve the quality of life and behavior of patients with cardiovascular diseases in low-resource settings, Islamabad, Pakistan.

Study Design Randomized controlled trial (RCTs) is the study and considered the appropriate level of studies that are evidence based and establish causal relationships in clinical research.

The applicability of this interventional study design is effective for prospective data collection, investigator-controlled intervention, usage of a concomitant control group, and randomizing to balance clear and latent confounding factors. Therefore, randomized controlled trial design will be more effective in this rigorous in improving positive outcomes of health by evaluating the effectiveness of home-based cardiac rehabilitation to improve the quality of life and behavior of the patients.

Study Setting The study will be conducted at the cardiac center of Pakistan Institute of Medical Sciences, Islamabad, which is a research-oriented health sciences institute located in Islamabad, Pakistan. It is one of the region's leading tertiary-level hospitals and teaching institutes, which includes both clinical and supporting services. It is almost a 1000-bed hospital that included medical, surgical, cardiac, gynecological, ENT, and burn care centers. PIMS hospital is the only hospital providing hospital based cardiac rehabilitation services to the population of Islamabad, Rawalpindi, Kashmir, and KPK.

The Cardiac Centre of the PIMS hospital is the only center in Islamabad among five tertiary hospitals that provides cardiac health services, including emergency medicine, surgical and diagnostic care, and operative cure and care. Therefore, the purpose of selecting this setting seemed to be appropriate for conducting this research study. Islamabad is the capital city of Pakistan and is located within the federal Islamabad Capital Territory. The population of this cosmopolitan city is more diverse and multi cultured.

Study Population Research Population The increased burden of CVD has become a serious health concern in Pakistan. Recent reports from Pakistan indicate higher rate of CVDs in the young population. Cardiovascular patients are assessed inaccurately, and their condition is misinterpreted resulting in appropriate medications leading to the older populations at the risk in cardiac management affecting their quality of life. Therefore, the patients more than 18 years age diagnosed with cardiovascular diseases based on diagnosis and clinical history including Electric Cardiogram, non-invasive tests like, echocardiography, exercise tolerance test (ETT), Thallium stress test, biochemical markers, and selected for procalcitonin PCI, a biomarker for the diagnosis of the infection in the heart. Patients discharged from the hospital by the consultant will be included for the research study.

Sample Size Calculation Sample size calculation is instrumental at the planning phase which make sure that there are sufficient and appropriate number of samples for provision of the reliable and accurate assessment of the drug items with certain statistical assurance. The purpose of sample size estimation is to plan sufficient figures of subjects for designed study design. Sample size planning is considered suitable strategy of calculating study subjects in mathematical manner of making a ballpark estimate. Sample size planning is considered essential for both analytic and descriptive study design, and the planning for estimation of sample size should earlier during the procedure of developing the research design so that appropriate modifications and can be made. Hence, the sample size is calculated on G Power software based on an expected moderate effect size of 0.59 to assess the effectiveness of home-based cardiac rehabilitation to improve the quality of life of cardiovascular patients in low- resource settings.

The following parameters were used for sample size calculation:

Assumptions:

* Effect size (Partial eta squared): 0.59
* Significance level (α): 0.05 (two-tailed)
* Power (1 - β): 0.80 (80%)
* Allocation ratio: 1:1 (equal participants in both groups)
* Dropout rate: 20%

The sample size per group is calculated using the following formula for comparing two independent means:

Therefore, the required sample size is approximately 46 participants per group (before adjusting for dropout).

To account for a 20% dropout rate:

Adjusted sample size per group = n / (1 - dropout rate) Adjusted n = 46 / (1 - 0.20) Adjusted n = 46 / 0.80 Adjusted n = 57.5 ≈ 58 participants per group Final total sample size = 58 (intervention) + 58 (control) = 116 participants Thus, a total of 116 participants (58 in each group) will be required to detect an effect size of 0.59 with 80% power and 5% significance level, accounting for a 20% dropout rate.

Randomization In clinical trials, statistical inference is a compulsory process to testify potency, efficacy and safety of drugs, procedures and medical devices, allowing generalization of the results observed through sampling process. Randomization is the allocation technique applied for study participants to study groups by chance Participants will be randomly assigned to either the hone based cardiac rehabilitation group or to the control group of routine/ standard care using a computer-generated sequence. Simple randomization can be adopted using technique of sealed envelopes during the sampling process. This strategy consists of a group assignment (with a new envelope being opened on enrollment of as each patient), or application of randomization software for randomization process. However, there is rare usage of sealed envelopes considering potential risks for investigator manipulation (Piantadosi, 2024). For instance, chronological bias, which cannot be ignored if there was recruitment of the study participants mismatched, and one group recruited earlier in the control group and/or the majority of those in the treatment group were recruited later. Restrictive randomization technique is effective to resolve the imbalance in simple randomization This simple strategy of randomization is suggested for large sample size in large-scale clinical trial studies because the possibility of imbalance in trials with a small number of samples is higher. Blocking is one of the effective strategies employed in the RCTs. In short block randomization is a technique that ensures that there is relatively equal number of study participants in each cohort. Block randomization has the advantage, which increases comparability between two groups by keeping the ratio of the number of study participants between cohorts almost similar. Therefore, the permuted- block randomization sampling technique will be adopted in this study. Blocking is technique of restricted randomization that maintains balance between the two sets at the end of every block. Technique of sealed envelope will be applied to allocate each study participants into either usual care or cardiac rehabilitation.

Selection of Criteria Inclusion Criteria

The study participants who will be included in the study who have been:

* Diagnosed with coronary artery disease, myocardial infarction and heart failure
* Diagnosed with cardiovascular diseases based on clinical history and diagnosis, including electrocardiogram (ECG), biochemical markers, or non-invasive tests like, echocardiography, exercise tolerance test (ETT), Thallium stress test, and selected for procalcitonin PCI, a biomarker for the diagnosis of the infection
* Either gender included
* Found medically stable and discharged from the hospital.
* Showed participation willingly and signed informed consent form
* Accessible to mobile phone communication or any other source of communication
* Resident of the surrounding areas other than the sectors of Islamabad as defined by the Capital Development Authority (CDA) of Pakistan.

Exclusion Criteria:

* Patients who have been diagnosed with comorbidity of psychiatric disorder or cognitive impairment
* Individuals with specific cardiac conditions or treatments, such as heart valve replacement, heart failure, or atrial fibrillation, or those with implanted cardiac devices like CRT or ICD.

Randomization and Allocation Participants will be randomly assigned to Intervention Group (HBCR): Will receive a structured home-based cardiac rehabilitation program.

Control Group: Will receive standard post-discharge care with routine follow-up.

Study Instrument Questionnaire 1 (Mac New Quality of Life Questionnaire) Self-reported questionnaire plays an essential role to assess quality of life using in a way to explore and evaluate psychological experience of participants with cardiac issues. Data gathered through the standardized and pre-tested Mac New Quality of Life questionnaire, which is a diagnostic instrument consisted of multiple-choice questions (MCQs). The MacNew Health-Related Quality of Life Questionnaire is an exponentially adopted instrument for the evaluation of health-related quality of life in cardiovascular patients. The validity and reliability and validity of the Italian version of the MacNew Questionnaire was determined in patients with angina, cardiac patients, such as myocardial infarction, angina or ischemic heart failure. The Italian Mac New version demonstrates There is a high internal consistency and reliability of the Italian Mac New version as per research studies (Cronbach's α ≥ 0.86). The Italian version of the Mac New Questionnaire shows higher satisfaction rate of psychometric properties with reliability and validity with heart failure, angina and MI. The Italian version of the Mac New Quality of Life questionnaire is comprised of 27 questions, included seven questions about clinical manifestations in three subscales that assess emotional, physical and social functions; a global health-related quality of life (HRQL) score is calculated from all scored sections. Study participants are directed to assess only one out of seven possible answers, each marked with a checkbox, and are not able to choose more than one answer for each proposed question for calculation of the last score. McNew is an exemplary successful and cognitive instrument that is immediately applicable and effective to evaluate the problems of cardiovascular (CVD) patients. This questionnaire has been used successfully in cardiac rehabilitation program studies. The Mac New Quality of Life after diagnostic evaluation of cardiovascular disease (Mac New QL) index includes 27 questions, with each having 7 optional response. The range of this questionnaire is 1.0 to 7.0, and the scoring scale comprises a 7-point Likert scale from a lower score of 1 to a higher score 7 as high quality score. There are both versions of Urdu and English with a worldwide score calculated as the average over all items.

3.4.2 Questionnaire (The Health Promoting Lifestyle Profile II (HPLP-II) The Health Promoting Lifestyle Profile II (HPLP-II) questionnaire is the updated version of the HPLP questionnaire and was developed first by Walker et al. HPLP-II questionnaire consisted of 52 items and the six-point subscale items for HPB. Questionnaire is available into multiple languages, such as Spanish, Japanese, Arabic, Chinese and Turkish, and its validity and reliability have been checked and verified. HPLP-II is a comprehensive instrument and tool for evaluating health behaviors of cardiovascular patients (Bermeo et al., 2024). Moreover, it is paramount to the evaluate of the intervention's effectiveness ratio in scientific studies associated elderly population. Whereas the Pakistan's population is aging Fastly and there are no effective study research instruments to evaluate health behaviors in elderly population. Therefore, it is essential that HPLP-II questionnaire is regionally localized as applied in Iranian population to assess the lifestyle of the adults and evaluate HPB. Researchers computed a significant concurrent validity (r = 0.63), and very high reliability (α = 0.98) of HPLP-II in Srilanka. Also, the validity and reliability of the HPL II questionnaire were examined in the Iranian research study. Additionally, the demographic variables in the (HPLP-II, the main questionnaire adopted in this research consisted updated version of the health-promoting lifestyle profile (HPLP-II) developed by Walker et al. first, and which has been made reliable and valid in the research study conducted by Zaidi et al. for Iranian elderly (under 60 years) population. The original version of this instrument comprises of 52 items that measure and evaluate HPB in six subscales (nutrition, physical activity, health responsibility, stress management interpersonal relationships, and spiritual growth). Each subscale consists of multiple subsections included as nutrition: Nine items; physical activity: Eight; health responsibility: Nine, stress management: Eight, interpersonal relationships: Nine; and spiritual growth: Nine. The choices for the questions are mentioned on a four-point Likert scale (never, sometimes, often, and routinely). Overall, the score for health-promoting lifestyle and behavioral areas is computed by using the mean of answers for all 52 items and for each subscale (eight or nine items) In this questionnaire 52 is the lowest and 208 is the highest total score, respectively. Item based total correlations were computed to measure the method of items of a scale differentiated the adults with regard to their HPB.

Next, to determine the internal consistency, Cronbach's alpha coefficient was used to determine the internal consistency, and to check the time reliability, the test-retest method was adopted Correlation between the scores was achieved from the two investigations during the duration of 2 weeks interval assessed by measuring the class correlation coefficient (ICC). Accepted values for Cronbach's alpha coefficient and ICC 0.7 are preferred more in the scientific studies Health Promoting Lifestyle Profile-II (HPLP-II) designed by Walker, Kerr, and Penderin 1990 were applied in the research studies. HPLP-II was translated SWBS in Urdu using Brislin translation method15 which included 20 items. Each item was designed to score on a 6- point rating scale ranged from strongly agree (1) to strongly disagree (6). Items 1, 2, 5, 6, 9, 12, 13, 16,, and Urdu version of the questionnaire showed moderately high reliability (α = 0.86). To assess health promoting lifestyle HPLP- II (52 items), 14 was applied in the study conducted in Pakistan (Sultan et al., 2022). Every item scored from 1 (Never) to 4 (Routinely) and composite high score showed positive outcome of health lifestyle. In this study, Urdu version of HPLP-II also showed high reliability.

Data Collection Method Data will be collected from the cardiology center of PIMS hospital after patients are diagnosed with cardiovascular disease by a cardiologist, and study participants will be recruited from the cardiology ward. Data will be collected at two points: baseline (preintervention within one week of enrollment in the study) and post-intervention (after the twelve weeks). Initially, baseline data will be collected, and the patients will then be randomized into usual care or a cardiac rehabilitation group. The cardiology center contains components such as a cardiology ward, cardiac surgery ward, coronary care unit, and cardiac emergency unit. A formal meeting will be held with the head nurse or nurse manager of the cardiac center. The head nurse will be informed about the purpose of the study, and the data collection procedure will be explained. Besides, IRB letters will be provided to them regarding approval and permission to conduct the research study. Patients' data will be collected from the cardiac center following the inclusion and exclusion criteria applicable to the study participants. Then informed consent will be given to the study participants who will show willingness to participate in their study. The informed consent attached in the annexure will contain details of the purpose, procedure, and ethical considerations of maintaining the anonymity, confidentiality, and privacy of the data and the option to withdraw from the study.

During the initial phase, the demographic and baseline data will be collected, such as name, gender, educational level, age, economic status, and marital status, from the study participants. Then data of clinical features such as smoking, Body Mass Index (BMI), and diagnosis with cardiovascular diseases. Moreover, researchers will collect the data of cardiac risk factors of included study participants. The data will contain blood pressure, heart rate, and other cardiac health-related clinical features. Besides, the patient's cognitive abilities and performance and motivation for behavioral changes will be assessed by the researcher. In the second phase, the researcher will examine functional capability, physical mobility and exercise, risk-factor modification, smoking cessation, medication adherence, nutritional guidance, and psychotherapy.

For qualifying this phase, an exercise test of 6-MWT will be conducted also. Additionally, a structured and developed copy of the HBCR will be shared with the study participants, and the contents of the copy will comprise physical mobility and exercise, methods for risk-factor change, dietary guidelines, and medication adherence guidelines and their importance. Similarly, the audiovisual material will be provided to the study participation regarding contents included in the HBCR guide, and this will continue from the first week to the 12th week.

The control group will receive only standard communication from the cardiologist and routine follow-up care. The control group will receive standard discharge advice and routine outpatient follow-up care as per hospital protocol, with no structured rehabilitation support. Home-based cardiac rehabilitation for the intervention group will be supervised by a multidisciplinary team such as a researcher, trained nursing staff, and cardiologist. A structured cardiac rehabilitation program will be conducted at the patient's home. This structured program will include dietary counseling, physical activity suggestions and recommendations, adherence to medications prescribed by the cardiologist, psychotherapy, and lastly telephone calls or visits at home. The time duration of the data collection will start from the baseline to the intervention, comprising 12 weeks.

Description of Variables

This quantitative study applies RCT research design to evaluate the effectiveness of homebased cardiac rehabilitation in low-resource settings. This study includes the two types of variables, which are the following:

Independent Variable Home-based cardiac rehabilitation is an independent and categorical variable in this study, which is a structured cardiac rehabilitation program, to evaluate the effectiveness of home-based cardiac rehabilitation.

Dependent Variables Quality of Life: It is a dependent and continuous variable, which will be evaluated from the study participants through a validated and reliable McNew Questionnaire containing three subdomains, such as physical, social, and emotional functioning. The scoring range starts from 1 to 07, whereas a high score indicates better quality of life. Time duration of measurement starting from baseline to the intervention comprising 12 weeks.

Health Behavior: It is a dependent and continuous variable, which will be evaluated from the study participants through a validated and reliable Health-Promoting Lifestyle Profile II (HPLP II) questionnaire containing three subdomains, such as diet, physical activity, medication adherence, smoking cessation, and stress management. Its scoring range is based on the Likert-type scale, such as 1 = never to 4 =, whereas a high score represents more quality behavior.

Outcome Measures Primary Outcome Quality of life Quality of life will be measured using validated tools such as the MacNew Quality of Life Questionnaire (description provided in study instrument section). Health Behavior Change Assessed using a self-reported questionnaire covering physical activity, diet, medication adherence, and smoking. Its scoring range is based on the Likert-type scale, such as 1 = never to 4 =, whereas a high score represents more quality behavior.

Secondary Outcome Frequency of Emergency Hospital Visits The frequency of emergency hospital visits will be recorded from the study participants till the till the 12th week of data collection and intervention.

Bio-Physiological Parameters Data of biophysiological parameters such as systolic and diastolic BP, heart rate, blood glucose, body mass index, LDL, high-density lipoprotein, triglyceride, and hemoglobin will be collected to assess physiological patterns affecting cardiac health.

Data Analysis Data will be analyzed using SPSS, updated version 25. Descriptive statistics such as mean and standard deviation will be calculated for continuous variables to evaluate characteristics of study participants. Percentages and frequencies will be presented for categorical variables. The ShapiroWilk normality test will be applied to evaluate the normality data, knowing that all variables had a p value of more than 0.05 to highlight parametric data. Besides, an independent sample test will be applied to compare the outcomes between the two groups. In this research study, a p-value lower that 0.05 will be considered statistically significant to evaluate the effectiveness of home-based cardiac rehabilitation program compared to the usual group of standard care.

Data Management Plan For managing data, codes will be allotted to each study participant. Different codes will be marked and labeled with either numbers or letters for recognition purposes. The primary researcher will maintain the proper documentation record of the study participants in the computer system. Proper procedure will be adopted for consistency and completeness of the record. The Epi data software version 3.1 will be utilized for the data entry purpose, and double entry data will be out by any expert data analyst and computer operator having vast experience in managing quantitative data of research studies. Consistencies of the data will be double-checked. After the double entry, two Data sets will be compared in terms of consistency for any missing data otherwise, correction will be made if an error is found before transferring data into the SPSS updated version 23 for data analysis.

Ethical Consideration:

Ethical approval will be obtained from the Institutional Review Board (IRB). A permission letter from an institution will be obtained. Written informed consent will be taken from all participants. Participants can withdraw at any point without any consequences. Data confidentiality and privacy will be strictly maintained.

ELIGIBILITY:
Inclusion Criteria:

Diagnosed with coronary artery disease, myocardial infarction and heart failure Diagnosed with cardiovascular diseases based on clinical history and diagnosis, including electrocardiogram (ECG), biochemical markers, or non-invasive tests like, echocardiography, exercise tolerance test (ETT), Thallium stress test, and selected for procalcitonin PCI, a biomarker for the diagnosis of the infection Either gender included Found medically stable and discharged from the hospital. Resident of the surrounding areas other than the sectors of Islamabad as defined by the Capital Development Authority (CDA) of Pakistan.

-

Exclusion Criteria:

-

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 92 (Estimated)
Dates: Start 2025-12-15 (Estimated); Primary Completion 2026-01-01 (Estimated); Study Completion 2026-03-15 (Estimated)

PRIMARY OUTCOMES:
Quality of life Questionnaire | Three months
  Quality of life Quality of life will be measured using validated tools such as the MacNew Quality of Life Questionnaire (description provided in study instrument section).
Health Behavior Change questionnaire | Three months
  Health Behavior Change Assessed using a self-reported questionnaire covering physical activity, diet, medication adherence, and smoking. Its scoring range is based on the Likert-type scale, such as 1 = never to 4 =, whereas a high score represents more quality behavior.

CONTACTS AND LOCATIONS:
Locations (1):
- Cardiac Centre Pakistan Institute of Medical Sciences Islamabad, Islamabad, Pakistan

IPD SHARING:
Plan to Share IPD: No